CLINICAL TRIAL: NCT04015167
Title: A Post-Market Clinical Evaluation of the Treatment of Tibia Fractures With the T2 Alpha Tibia Nailing System
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: T2 Alpha Tibia
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- T2 Alpha Tibia: Subjects in the clinical investigation will undergo placement of the Tibial Nail of the T2 Alpha Tibia Nailing System, according to the approved Instructions for Use and Operative Technique Manual.
  Interventions: Device: T2 Alpha Tibia Nailing System

INTERVENTIONS:
Device: T2 Alpha Tibia Nailing System — The T2 Alpha Tibia Nailing System is intended for temporary stabilization of bone segments or fragments until bone consolidation has been achieved.

SUMMARY:
This investigation is a prospective, multi-center clinical investigation. It is anticipated that a total of 80 subjects will be enrolled. Neither subjects nor investigators are blinded to treatment and the clinical investigation includes a historical control which will be compared to the T2 Alpha Tibia Nailing System.

Total duration of enrollment, 12 month follow-up and analysis is expected to take 31 months. The clinical investigation has been designed to follow the surgeon's standard of care for tibia fractured subjects, in addition to a 12 month follow-up visit.

The primary endpoint of this clinical investigation is to confirm efficacy/performance at 12 months, as measured by the SF-36 Physical Component Summary (PCS). Confirmation of efficacy/performance at 12 months will be based on an equal or higher (non-inferior) SF-36 Physical Component Summary (PCS) result of the T2 Alpha Tibia Nailing System compared to the benchmark literature.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the T2 Alpha Tibia Nailing System. Efficacy/performance of the procedure will be measured by an equal or higher (non-inferior) SF-36 Physical Component Summary (PCS) score result of the T2 Alpha Tibia Nailing System compared to the T2 Tibia benchmark literature at 12 months.

In addition, demonstration of bone consolidation in correct alignment will be measured by Investigator assessment by 12 months. Safety of the T2 Alpha Tibia Nailing System will be demonstrated through reporting of device related intra-operative and post-operative Adverse Events/incidents by 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female age 18 years or older at the time of surgery;
* Subject is willing and able to give written informed consent and comply with the requirements of this Clinical Investigation Plan;
* Subject is intended to be, treated with the Tibial Nail of the T2 Alpha Tibia Nailing System in accordance with the following legally cleared/ approved Indications for Use:

Indications for Use approved In United States and Canada include:

* Open and closed tibial fractures
* Pseudoarthrosis and correction osteotomy
* Pathologic fractures, impending pathologic fractures and tumor resections
* Fractures involving osteopenic and osteoporotic bone
* Nonunions and malunions

Exclusion Criteria:

* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device clinical investigation that, in the opinion of the Investigator, may confound results;
* Per the Investigator, the subject is in poor general health or undergoing any concurrent disease that would place the subject in excessive risk to surgery (i.e. significant circulatory problems, cardiac disease).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 80 subjects are to be enrolled in this clinical investigation. Subjects participating in this clinical investigation will be recruited from the investigator's standard subject population, where all subjects presenting for treatment of tibial fractures will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (4):
- United States (4):
  - St. Cloud Orthopedic Associates, Ltd, Sartell, Minnesota
  - New York University, New York, New York
  - UC Health, Cincinnati, Ohio
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2 Alpha Tibia
Started | 103
Completed | 55
Not Completed | 48
Not completed — Lost to Follow-up | 40
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 2
Not completed — Subject went to jail | 1

BASELINE CHARACTERISTICS:
Arm/Group | T2 Alpha Tibia
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.81 (18.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 5
  Ethnicity: Black or African | 26
  Ethnicity: Caucasian | 72
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: SF-36 PCS (36-Item Short Form Health Survey Physical Component Summary)
Description: The primary endpoint of this clinical investigation is to confirm efficacy/performance at 12 months, as measured by the SF-36 PCS (36-Item Short Form Health Survey Physical Component Summary). The SF-36 PCS is a self-report measure of health status. SF-36 Physical Component Summary scores range from 0 to 100; higher SF-36 score results are linked to better subject results.
  Confirmation of efficacy/performance at 12 months will be based on an equal or higher (non-inferior) SF-36 Physical Component Summary (PCS) result of the T2 Alpha Tibia Nailing System compared to the T2 Tibia benchmark literature.
Time Frame: 12 months
Population: Of the 55 subjects that completed the study, 53 subjects were available for the SF-36 assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T2 Alpha Tibia
Number analyzed (Participants) | 53
score on a scale | 49.21 (9.65)

2. Secondary Outcome: Safety Will be Measured by Capturing the Incidence Rate of Device-related Adverse Events
Description: Incidence of device-related adverse events will be monitored by 12 months through data collection and analyses.
Time Frame: 12 months
Population: 11 out of 103 subjects had reportable Adverse Events.
Measure: Count of Participants; unit: Participants
Arm/Group | T2 Alpha Tibia
Number analyzed (Participants) | 11
Participants
  *Delayed union (no bone consolidation within 4 months) | 2
  Implant loosening (screw) | 1
  Infection (deep) | 2
  Non-union (no bone consolidation within 6 months) | 2
  Pain | 4

3. Secondary Outcome: Efficacy/Performance Will be Measured by Demonstration of Bone Consolidation
Description: Bone consolidation will be assessed by 12 months as measured by Investigator assessment.
Time Frame: 12 months
Population: of the 55 subjects that completed the study, 54 subjects were available for bone consolidation assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | T2 Alpha Tibia
Number analyzed (Participants) | 54
Participants
  Bone Consolidation - Yes | 48
  Bone Consolidation - No | 6

ADVERSE EVENTS:
Time Frame: 1 year
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | T2 Alpha Tibia
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 11/103
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T2 Alpha Tibia (N=103)
Delayed union (no bone consolidation within 4 months) (Musculoskeletal and connective tissue disorders) | 2
Implant loosening (screw) (Product Issues) | 1
Infection (deep) (Infections and infestations) | 2
Non-union (no bone consolidation within 6 months) (Musculoskeletal and connective tissue disorders) | 2
Pain (Product Issues) | 4

LIMITATIONS AND CAVEATS:
Assessment of long-term impacts were challenging due to a higher number of loss-to-follow-up, which resulted in missing data and reduced statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04015167/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04015167/SAP_001.pdf